CLINICAL TRIAL: NCT04627155
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Human Tolerance and Kinetics of LY03003 By Single Intramuscular Injection
Brief Title: A Study to Evaluate the Human Tolerance and Pharmacokinetics of LY03003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03003/CT-CHN-101
Record Dates: First submitted 2020-11-05; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Parkinson Disease
Keywords: LY03003
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7mg dose group (Experimental)
  Interventions: Drug: LY03003
- 14mg dose group (Experimental)
  Interventions: Drug: LY03003

INTERVENTIONS:
Drug: LY03003 — Rotigotine,extended-release microspheres

SUMMARY:
This study is to evaluate the human tolerance and pharmacokinetics of LY03003.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 to 45 years, no less than one-third of a single sex ratio;
2. normal physical examination items (including general physical examination, blood and urine, blood biochemistry, anti-HBV, anti-HCV, anti-HIV, pregnancy test, ECG, chest X-ray);
3. body weight not less than 50 kg, body mass index between 19 and 24 kg/m2;
4. during 2 weeks not using any drugs;
5. no history of drug allergy or drug allergy;
6. voluntarily participate in this clinical trial, can cooperate to complete the specified examinations, and sign the informed consent form

Exclusion Criteria:

1. abnormal health examination and clinical significance;
2. history of allergy to non-ergot dopamine agonists, or history of allergy to other drugs and food;
3. Bronchial asthma, epilepsy, mechanical intestinal obstruction, urinary tract obstruction;
4. history of liver and kidney disease, cardiovascular system, respiratory system, hematopoietic system, nervous and mental illness;
5. Women of childbearing age who have a positive pregnancy test or a negative pregnancy test but cannot ensure to take appropriate contraceptive measures during the study;
6. lactating women;
7. Male subjects who are unwilling to take appropriate contraceptive measures. Appropriate measures include the use of condoms, spermicides, or female partners using intrauterine devices (IUDs), ovarian caps, oral contraceptives, injected or subcutaneously implanted progestins, and tubal ligation surgery. Female partners must not be pregnant or lactating women;
8. smokers, alcoholics and drug abusers;
9. drinkers within 24 hours before medication;
10. used any drugs within 2 weeks before the trial; Use of drugs with effect on liver and kidney function within 11.3 months; Participated in other drug trials within 12.3 months, donated blood loss (≥ 200ml), or sampled as subjects;

13. Researchers believe that the participants are not suitable.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2013-05-20 (Actual); Study Completion 2013-05-20 (Actual)

PRIMARY OUTCOMES:
Plasma drug concentration | Hour1 、Hour6、Hour12、Hour24、Hour36、Hour48、Hour60 、Hour72 、Hour84、Hour96 、Hour120 、Hour144 、Day8、Day9、Day10、Day11、Day12、Day13、Day14、Day16、Day18 and Day 21after injection
  Cmax

SECONDARY OUTCOMES:
Vital signs | Hour1 、Hour6、Hour12、Hour24、Hour36、Hour48、Hour60 、Hour72 、Hour84、Hour96 、Hour120 、Hour144 、Day8、Day9、Day10、Day11、Day12、Day13、Day14、Day16、Day18 and Day 21after injection
  Blood pressure
Vital signs | Hour1 、Hour6、Hour12、Hour24、Hour36、Hour48、Hour60 、Hour72 、Hour84、Hour96 、Hour120 、Hour144 、Day8、Day9、Day10、Day11、Day12、Day13、Day14、Day16、Day18 and Day 21after injection
  Weight